CLINICAL TRIAL: NCT06118593
Title: Why in Hospital After ERAS VATS Wedge Resection
Brief Title: Why in Hospital After Wedge Resection
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lin Huang, Department of Cardiothoracic Surgery, Rigshospitalet, Denmark
Other Study IDs: P-2022-238
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Thoracic Surgery, Video-Assisted; Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the realm of lung surgery, video-assisted thoracoscopic surgery (VATS) offers distinct advantages, including shorter hospital stays, reduced pain, improved quality of life, and increased postoperative mobility when compared to thoracotomy. Additionally, the enhanced recovery after surgery (ERAS) protocol in lung surgery, characterized by a comprehensive, multidisciplinary approach, have streamlined postoperative recovery, resulting in early discharge and diminished postoperative complications. However, drawing from our extensive experience with fully implemented ERAS VATS for patients undergoing pulmonary lobectomy, we observed that approximately 45% of patients did not experience early discharge.

Based on existing evidence, the length of stay (LOS) following wedge resection typically ranges from 3 to 6 days across various regions, including Europe, the United States, and China. However, there is a notable lack of procedure-specific data for ERAS VATS wedge resection to explore reasons of delaying discharge. This prompts us to undertake an investigation into individuals following pulmonary wedge resection under the same ERAS programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent video-assisted thoracoscopic surgery wedge resection

Exclusion Criteria:

* < 18 year old
* Unable to understand Danish
* No residence in the Eastern Denmark
* Transfer to anatomical resection or cancel surgery
* Reject to join or withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent video-assisted thoracoscopic surgery wedge resection.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Length of stay | Up to the day of discharge
  Number of overnight stay
Reasons for staying in hospital | Up to the day of discharge
  patient-reported outcomes for why in hospital, including pain or social factors; postoperative complications, diagnosed by clinicians

SECONDARY OUTCOMES:
Postoperative pain scale | At the day of surgery
  The pain scale (from 0 to 10) will be evaluated by patients.
Duration of chest drain | Up to the day of chest drain removed
  Days of chest drain placed
Postoperative complications | Up to postoperative day 30
  Diagonosis is following ICD-10
30-day readmissions | Up to postoperative day 30
  Admission to hospital again within 30 days after surgery
Postoperative activity | At the day of surgery
  Patients report whether they can stand up, walk within 6 meters, or walk over 6 meters, up to 3 and 6 hours after surgery
Opioid usage | At the day of surgery and at the day of discharge
  It is classified as opioid used and no opioid used

CONTACTS AND LOCATIONS:
Overall Officials: René H Petersen, Study Director — Department of Cardiothoracic Surgery, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The data is possible shared to other researchers if they contact with study director and the approvals are obtained subsequently.

REFERENCES:
- [Derived] Huang L, Kehlet H, Petersen RH. Why do patients stay in hospital after enhanced recovery thoracoscopic wedge resection? A prospective observational study. Eur J Cardiothorac Surg. 2024 Oct 1;66(4):ezae366. doi: 10.1093/ejcts/ezae366. PMID 39374548